CLINICAL TRIAL: NCT04353128
Title: Multicenter Randomized Controlled Trial of the Efficacy of Melatonin in the Prophylaxis of SARS-coronavirus-2 Infection Among High Risk Contacts.
Brief Title: Efficacy of Melatonin in the Prophylaxis of Coronavirus Disease 2019 (COVID-19) Among Healthcare Workers.
Acronym: MeCOVID
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MeCOVID
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2020-04

CONDITIONS: Covid19; SARS-CoV 2; Coronavirus Infection
Keywords: melatonin; prevention; covid19; Sars-CoV2; healthcare
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): 2 mg of melatonin orally before bedtime for 12 weeks
  Interventions: Drug: Melatonin 2mg
- Placebo (Placebo Comparator): Identically looking placebo orally before bedtime for 12 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Melatonin 2mg — 2 mg of prolonged release melatonin tablets per os (P.O.) before bedtime for 12 weeks
  Other Names: circadin 2 mg
  Arms: Melatonin
Drug: Placebo oral tablet — Identically looking placebo tablets P.O. before bedtime for 12 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
There is an urgent need to evaluate interventions that can prevent the infection with SARS-CoV 2 of healthcare workers at risk. Melatonin is an inexpensive and safe product with protective effect in both bacterial and viral infections likely due to its anti-inflammatory and anti-oxidative effects. This randomized controlled trial seeks to evaluate is efficacy as a prophylaxis in healthcare workers exposed to the virus in their clinical practice.

DETAILED DESCRIPTION:
Healthcare workers are at an increased risk of acquiring COVID-19 due to an increased exposure to the virus and global personal protective equipment shortages. Preventing the infection of healthcare workers is critical the current epidemic situation when healthcare systems are under extreme pressure. There is a lack of evidence surrounding potential preventive strategies to decrease the incidence of COVID-19 among healthcare workers.

Melatonin, an endogenous hormone involved in circadian rhythm control, is an inexpensive and safe product that has shown protective effects in bacterial and viral infections likely due to its anti-inflammatory and anti-oxidative effects.

SARS-CoV 2 seems to relatively spare younger children and those who are infected develop the severe forms of the disease very rarely. Peak melatonin serum levels are higher in younger children and decrease with age. These levels are also higher in women, specially during pregnancy, who also seem to be less affected by the virus when compared to men.

The investigators hypothesize that elevating peak melatonin levels to a range similar to that of children by administering 2 mg of melatonin daily might prevent the infection with SARS-CoV 2 among exposed healthcare workers. The investigators also hypothesize that among those who develop the disease melatonin might prevent the more severe forms.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers from the public and private Spanish hospital network at risk of SARS-CoV 2 infection
* Not having a previous COVID19 diagnosis
* Not having experienced COVID19 symptoms from March 1st 2020 until randomization
* Understanding the purpose of the trial and not having taken any pre-exposure prophylaxis (PrEP) including HIV PrEP from March 1st 2020 until randomization
* Having a negative SARS-CoV 2 CRP before randomization
* Having a negative urinary pregnancy test in the previous 7 days for premenopausal women
* Premenopausal women and males with premenopausal couples must commit to using a high efficiency anticonceptive method

Exclusion Criteria:

* HIV infection
* Active hepatitis B infection
* Renal failure (CrCl < 60 mL/min/1.73 m2) or need for hemodialysis
* Osteoporosis
* Myasthenia gravis
* Retinitis pigmentosa
* Bradycardia (less than 50 bpm)
* Weight less than 40 Kg
* Treatment with drugs that prolong the QT interval for more than 7 days in the last month before randomization including: azithromycin, cisapride, methadone, droperidol, sotalol, quinidine, clarithromycin, haloperidol...
* Hereditary intolerance to galactose, Lapp lactase deficiency or glucose or galactose malabsorption
* Treatment with fluvoxamine
* Treatment with benzodiazepines or benzodiazepine analogues such as zolpidem, zopiclone or zaleplon
* Pregnancy
* Breastfeeding
* History of potentially immune derived diseases such as: lupus, Crohn's disease, ulcerative colitis, vasculitis or rheumatoid arthritis
* Insulin-dependent diabetes mellitus
* Known history of hypersensitivity to the study drug or any of its components
* Patients that should not be included in the study at the judgment of the research team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
SARS-CoV 2 infection rate | up to 12 weeks
  Number of confirmed (positive CRP) symptomatic infections in each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Pedro de la Oliva, MD, PhD, Study Chair — Hospital Universitario La Paz; Antonio J Carcas, Study Chair — Hospital Universitario La Paz; Irene García García, Study Chair — Hospital Universitario La Paz; Amelia Rodríguez Mariblanca, Study Chair — Hospital Universitario La Paz; Lucía Martínez de Soto, Study Chair — Hospital Universitario La Paz; María J Rosales, Study Chair — Hospital Universitario La Paz; José R Arribas, Study Chair — Hospital Universitario La Paz; Juan González, Study Chair — Hospital Universitario La Paz; Alberto M Borobia, MD, PhD, Study Chair — Hospital Universitario La Paz; Miguel Rodriguez-Rubio, MD, Study Chair — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee PI, Hu YL, Chen PY, Huang YC, Hsueh PR. Are children less susceptible to COVID-19? J Microbiol Immunol Infect. 2020 Jun;53(3):371-372. doi: 10.1016/j.jmii.2020.02.011. Epub 2020 Feb 25. No abstract available. PMID 32147409
- [Background] Lu X, Zhang L, Du H, Zhang J, Li YY, Qu J, Zhang W, Wang Y, Bao S, Li Y, Wu C, Liu H, Liu D, Shao J, Peng X, Yang Y, Liu Z, Xiang Y, Zhang F, Silva RM, Pinkerton KE, Shen K, Xiao H, Xu S, Wong GWK; Chinese Pediatric Novel Coronavirus Study Team. SARS-CoV-2 Infection in Children. N Engl J Med. 2020 Apr 23;382(17):1663-1665. doi: 10.1056/NEJMc2005073. Epub 2020 Mar 18. No abstract available. PMID 32187458
- [Background] Scholtens RM, van Munster BC, van Kempen MF, de Rooij SE. Physiological melatonin levels in healthy older people: A systematic review. J Psychosom Res. 2016 Jul;86:20-7. doi: 10.1016/j.jpsychores.2016.05.005. Epub 2016 May 10. PMID 27302542
- [Background] Gunn PJ, Middleton B, Davies SK, Revell VL, Skene DJ. Sex differences in the circadian profiles of melatonin and cortisol in plasma and urine matrices under constant routine conditions. Chronobiol Int. 2016;33(1):39-50. doi: 10.3109/07420528.2015.1112396. Epub 2016 Jan 5. PMID 26731571
- [Background] Zhang R, Wang X, Ni L, Di X, Ma B, Niu S, Liu C, Reiter RJ. COVID-19: Melatonin as a potential adjuvant treatment. Life Sci. 2020 Jun 1;250:117583. doi: 10.1016/j.lfs.2020.117583. Epub 2020 Mar 23. PMID 32217117
- [Background] Tan DX, Korkmaz A, Reiter RJ, Manchester LC. Ebola virus disease: potential use of melatonin as a treatment. J Pineal Res. 2014 Nov;57(4):381-4. doi: 10.1111/jpi.12186. Epub 2014 Oct 14. PMID 25262626
- [Background] Ran L, Chen X, Wang Y, Wu W, Zhang L, Tan X. Risk Factors of Healthcare Workers With Coronavirus Disease 2019: A Retrospective Cohort Study in a Designated Hospital of Wuhan in China. Clin Infect Dis. 2020 Nov 19;71(16):2218-2221. doi: 10.1093/cid/ciaa287. PMID 32179890
- [Background] Gooneratne NS, Edwards AY, Zhou C, Cuellar N, Grandner MA, Barrett JS. Melatonin pharmacokinetics following two different oral surge-sustained release doses in older adults. J Pineal Res. 2012 May;52(4):437-45. doi: 10.1111/j.1600-079X.2011.00958.x. Epub 2012 Feb 21. PMID 22348451
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533